CLINICAL TRIAL: NCT03575169
Title: The Use of Bispectral Index Monitoring to Assess Depth of Sedation in Patients With Traumatic Brain Injury
Acronym: BIS-TBI
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1-063-18
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Traumatic Brain Injury
Keywords: Bispectral index; Monitoring; Sedation; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with TBI: Admitted to Aberdeen ICU with diagnosis of TBI and expected to require greater than 24 hours sedation.
  Interventions: Device: BIS Monitor

INTERVENTIONS:
Device: BIS Monitor — Unilateral BIS electrode

SUMMARY:
An observational study to assess the BIS reported level of sedation of patients with traumatic brain injury in the ICU.

DETAILED DESCRIPTION:
Patients admitted to Aberdeen ICU with severe traumatic brain injury will have a BIS electrode placed and observed for 24 hours. The study team will be blinded to the result, so not to influence treatment.

All clinical care is at the discretion of the clinical team.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18)
* Diagnosis of traumatic brain injury
* Expected to survive
* Expected to require greater than 24 hours of sedation and mechanical ventilation

Exclusion Criteria:

* Brain injury thought to be unsurvivable by ICU clinical team
* Frontal decompressive craniectomy
* Use of ketamine infusion at recruitment or planned use within 24 hours
* Fractured frontal bone or severe overlying soft tissue injury
* Simple extradural haemorrhage with no other obvious intracranial injury
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe traumatic brain injury requiring sedation and mechanical ventilation who are admitted to Aberdeen ICU.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mean BIS | 24 hours
  Mean BIS of patients sedated

SECONDARY OUTCOMES:
Mean ICP | 24 hours
  Mean ICP of sedated patient
Incidence of osmotherapy use | 24 hours
  Number of instances of osmotherapy use in sedated patients
Vasopressor dose | 24 hours
  Total vasopressor dose for sedated patients
Sedative dose | 24 hours
  Total sedative dose for sedated patients
Length of ICU stay | Days to weeks
  Number of days admitted to ICU

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Intensive Care Unit, Aberdeen Royal Infirmary, Aberdeen
  - NHS Tayside, Dundee
  - NHS Lothian, Edinburgh
  - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaye C, Rhodes J, Austin P, Casey M, Gould R, Sira J, Treweek S, MacLennan G. Assessment of depth of sedation using Bispectral Index monitoring in patients with severe traumatic brain injury in UK intensive care units. BJA Open. 2024 May 28;10:100287. doi: 10.1016/j.bjao.2024.100287. eCollection 2024 Jun. PMID 38868457